CLINICAL TRIAL: NCT03888625
Title: Randomized Clinical Trials to Compare the Healing Process of Idiopathic Macular Hole With Different Surgical Techniques
Brief Title: Compare the Healing Process of Idiopathic Macular Hole With Different Surgical Techniques
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Mauricio Maia, Professor of Ophthalmology Dept, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMH2019
Record Dates: First submitted 2019-03-21; First posted 2019-03-25 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Macular Holes
Keywords: macular holes
MeSH Terms: conditions — Retinal Perforations

STUDY DESIGN:
Intervention Model Description: In Group A, patients will undergo peeling with complete removal of the internal limiting membrane (ILM) and in the group B, the inverted ILM peeling technique will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Conventional ILM peeling (Active Comparator): peeling with complete removal of the internal limiting membrane (ILM)
  Interventions: Procedure: Conventional ILM Peeling
- GroupB: Inverted ILM Peeling (Active Comparator): the inverted ILM peeling technique, in which the ILM is left in the edge of the macular hole and the free area is inverted over the macular hole before fluid-air exchange
  Interventions: Procedure: Inverted ILM Peeling

INTERVENTIONS:
Procedure: Conventional ILM Peeling — peeling with complete removal of the internal limiting membrane (ILM)
  Arms: Group A: Conventional ILM peeling
Procedure: Inverted ILM Peeling — the inverted ILM peeling technique - the technique of Inverted flap described by Michalewska, in which the ILM is left in the edge of the macular hole and the free area is inverted over the macular hole before fluid-air exchange
  Arms: GroupB: Inverted ILM Peeling

SUMMARY:
To compare anatomic and functional results, and to evaluate postoperatively the healing process in 2 different techniques for the closure of the macular holes (MH)

DETAILED DESCRIPTION:
Patients with macular holes classified in stages 3 and 4 will be randomized into 2 groups. . In Group A, patients will undergo peeling with complete removal of the internal limiting membrane (ILM) and in the group B, the inverted ILM peeling technique will be performed. The 20% sulfur hexafluoride (SF6) gas will be used as a tamponade agent in all surgeries, and patients will be instructed to avoid the prone position for 5 days.

OCT images will be performed in the first 5 postoperative days and months 1, 3 and 6.

The primary outcome is anatomic closure of the MH closure in the month 6. The second outcomes are: mean best corrected visual acuity (BCVA) at month 6, mean change in the BCVA at month 6; integrity of the perifoveal external limiting membrane and ellipsoid zone on Optical Coherence Tomography (OCT); MH closure rate over time in days; functional improvement of microperimetry Statistical analysis will be performed with Student t-test and the p-value of ≤ 0.05 is considered significant.

ELIGIBILITY:
Inclusion Criteria:

> Stage 3 and 4 macular holes with visual acuity between 20/30 and 20/800 according to the ETDRS chart.

Exclusion Criteria:

* Macular holes secondary to ocular trauma, myopia or retinal detachment
* Any previous treatment for the macular hole
* Evidence on examination of any diabetic retinopathy
* History or presence of wet or dry age macular degeneration (AMD)
* Presence of epiretinal membrane or prior uveitis
* Any ocular surgery within 3 months before baseline
* Intra or periocular infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-06-15 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Anatomic closure | Month 6 post operative
  Rate of anatomic macular hole closure in the OCT at month 6

SECONDARY OUTCOMES:
BCVA mean | Month 6 post operative
  mean best corrected visual acuity (BCVA) at month 6
BCVA change | Screening and Month 6 post operative
  change in the BCVA at month 6
Integrity Membrane measured in microns (μm) by OCT | Month 6 post operative
  In the month 6, the area of discontinuity of the perifoveal external limiting membrane and ellipsoid zone in the OCT images will be measured in microns (μm) and correlated between groups

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Maia, MD, PhD, Study Director — Federal University of São Paulo
Locations (1):
- Dept. of Ophthalmology, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No